CLINICAL TRIAL: NCT05881577
Title: The Effect of Allergic Rhinitis on Educational Outcomes - a Register-based Study
Brief Title: The Effect of Allergic Rhinitis on Educational Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Ernst & Young (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI-X-06
Record Dates: First submitted 2023-02-16; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: The primary study population will consist of subjects with AR
  Interventions: Other: Observational
- Matched controls: children with no history of AR
- Sibling controls: siblings of the subjects in the case group with no history of AR

INTERVENTIONS:
Other: Observational — Impact of AR on educational outcomes
  Groups: Cases

SUMMARY:
The study will assess the the burden of living with allergic rhinitis (AR) and the effect of AR on school performance for children and adolescents in Denmark.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of AR on school performance and examination test grades for children and adolescents diagnosed with AR early in life, as well as analyse their burden of disease and healthcare resource use using real-world data from the exhaustive Danish population registers. This is a retrospective registry analysis that uses Danish registers during 1994 and 2021.

In Denmark, national registers collect data for the entire Danish population from birth to death and have done so for decades. This exhaustive data creates a sound foundation for this study of the impact of school performance caused by AR, as subjects can be traced with high certainty and detail over several years.

ELIGIBILITY:
Inclusion Criteria:

* The main study population (cases) consists of children who have been diagnosed with AR before turning 13. Diagnosis of AR will be identified by dispensations of prescribed AR medications, ICD-10 codes of AR-related hospitalisations and reimbursement codes for AR-related healthcare contacts in the primary healthcare sector.

At least two dispensed prescriptions of product containing intranasal corticosteroids (INCS) or antihistamines during the same calendar year for two consecutive years OR at least one visit with the primary healthcare sector with registered AR consultations AND at least one dispensed prescriptions of product containing INCS or antihistamines OR at least one contact with the hospital sector with an ICD-10 code for AR (primary or secondary diagnosis).

Exclusion Criteria:

* Children with their first AR-related healthcare contact or first AR-specific dispensed prescription at the age of 13 or older will be excluded.

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: children who have been diagnosed with AR before turning 13
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary school final examination test grades (oral and written) in: Language (Danish, English), Mathematics Obtained high school degree Obtained university degree | 1994-2021
  Test grades

SECONDARY OUTCOMES:
Cost of inpatient and outpatient hospitalisation | 1994-2021
  Cost in DKK
Cost of prescription medicine | 1994-2021
  Cost in DKK
Number of inpatient and outpatient visits | 1994-2021
  The number of inpatient/outpatients visits per year.

CONTACTS AND LOCATIONS:
Locations (1):
- ALK Abello, Hørsholm, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided